CLINICAL TRIAL: NCT04808284
Title: Neuromodulation in COVID-19 Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRJ2007
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; transcranial direct current stimulation (tDCS); executive function; depression; anxiety; autonomic nervous system; motor function
MeSH Terms: conditions — COVID-19; Depression; Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS-SMA (Experimental): Participants randomized to this arm will receive a single tDCS session delivered at 2mA to the supplementary motor area (SMA) for 30 minutes.
  Interventions: Device: Transcranial direct-current stimulation
- tDCS- DLPFC (Experimental): Participants randomized to this arm will receive a single tDCS session delivered at 2mA to the right (cathodal) and left (anodal) dorsolateral prefrontal cortex (DLPFC) for 30 minutes.
  Interventions: Device: Transcranial direct-current stimulation
- tDCS- SHAM (Sham Comparator): Participants randomized to this arm will receive a single session of Sham tDCS for 30 minutes, delivered to supplementary motor area (SMA) or to the right (cathodal) and left (anodal) dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Sham Transcranial direct-current stimulation

INTERVENTIONS:
Device: Transcranial direct-current stimulation — A single tDCS session will be delivered to the supplementary motor area (SMA) by a DC stimulator (NeuroConn, Germany). During stimulation, a pair of saline-soaked sponge electrodes (surface 35 cm²) will be used, with one electrode (anode) placed 1,8 cm forward Cz and the other electrode (cathode) over the right supraorbital region, according to the International 10-20 EEG system. Current intensity will be ramp up for 30 seconds until reaches 2 mA, and after 30 minutes current intensity will be ramp down for 30 seconds.
  Other Names: Active Transcranial direct-current stimulation; tDCS
  Arms: tDCS-SMA
Device: Transcranial direct-current stimulation — A single tDCS session will be applied bilaterally over the dorsolateral prefrontal cortex (DLPFC) by a DC stimulator (NeuroConn, Germany). During stimulation, a pair of saline-soaked sponge electrodes (surface 35 cm²) will be placed over F3 (anode) and F4 (cathode), according to the International 10-20 EEG system. Current intensity will be ramp up for 30 seconds until reaches 2 mA, and after 30 minutes current intensity will be ramp down for 30 seconds.
  Other Names: Active Transcranial direct-current stimulation; tDCS
  Arms: tDCS- DLPFC
Device: Sham Transcranial direct-current stimulation — A single Sham-tDCS session will be applied bilaterally over the dorsolateral prefrontal cortex (DLPFC) or over the supplementary motor area (SMA) by a DC stimulator (NeuroConn, Germany). A pair of saline-soaked sponge electrodes (surface 35 cm²) will be placed according to the International 10-20 EEG system. For SMA , one electrode (anode) will be placed 1,8 cm forward Cz and the other electrode (cathode) over the right supraorbital region. For DLPFC, electrodes will be placed over F3 (anode) and F4 (cathode). Current intensity will be ramp up for 30 seconds until reaches 2 mA, and after 30 seconds current intensity will be ramp down for 15 seconds.
  Other Names: Sham TDCS
  Arms: tDCS- SHAM

SUMMARY:
This clinical study is aimed at investigating the effects of transcranial direct current stimulation (tDCS) on COVID-19 patients not admitted to the intensive care unit. The tDCS is a non-invasive brain stimulation technique which applies a low intensity electrical current in order to modulate neuronal activity. Patients included will be submitted to a single session with active or sham tDCS, aiming to modulate prefrontal or supplementary motor area (SMA). Evaluation protocol will be performed before and after stimulation to verify the incidence of adverse events related to treatment and whether tDCS would affect measures of executive functioning, mood, anxiety, autonomic response and motor function in COVID-19 patients. We hypothesize the neuromodulation would be a safety, promising treatment to reduce possible impairments in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed diagnosis for SARS-CoV-2;
* ability to understand and execute the proposed protocol;
* vital signs (body temperature <38ºC, blood pressure between 90 x 60mmHg and 140 x 90 mmHg, respiratory rate between 12 e 30 bpm).

Exclusion Criteria:

* dyspnea or signs of respiratory effort;
* SpO2 ≤ 90%;
* hemodynamic instability;
* deep vein thrombosis, active bleeding, use of cardiac pacemaker;
* injury, pain or metallic implants in the cranium or scalp;
* seizure history;
* suspected or confirmed pregnancy;
* concomitant or previous rheumatic or neurological diseases;
* severe psychiatric diseases (schizophrenia, bipolar disorder, intellectual disability);
* severe musculoskeletal and/or integumentary disorders;
* severe psychiatric disorders;
* severe liver or kidney disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to treatment (safety) | post-treatment (up to one hour after the end of the treatment)
  Safety as assessed by incidence of adverse events by type, frequency, severity, and causality
Change from baseline autonomic response at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Heart rate variability (HRV) parameters change from pre-treatment to post-treatment
Change from baseline Trial Making Test (TMT) score at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Trial Making Test (TMT) score changes from pre-treatment to post-treatment
Change from baseline Digit span score at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Digit span score changes from pre-treatment to post-treatment
Change from baseline balance parameters at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Balance parameters change from pre-treatment to post-treatment
Change from baseline gait parameters at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Gait parameters change from pre-treatment to post-treatment

SECONDARY OUTCOMES:
Change from baseline Functional Status Score for the intensive care unit (FSS-ICU) at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Functional Status Score for the intensive care unit (FSS-ICU) changes from pre-treatment to post-treatment
Change from baseline Functional Reach Test (FRT) distances at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Maximum distances reached by subject change from pre-treatment to post-treatment
Change from baseline Beck Depression Inventory-II (BDI-II) score at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Beck Depression Inventory-II (BDI-II) score changes from pre-treatment to post-treatment
Change from baseline Beck Anxiety Inventory (BAI) score at the end of the treatment | pre-treatment (baseline), post-treatment (up to one hour after the end of the treatment)
  Beck Anxiety Inventory (BAI) score changes from pre-treatment to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda F Tovar-Moll, PhD, Study Director — D'Or Institute for Research and Education (IDOR); Erika C Rodrigues, PhD, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- D'Or Institute for Research and Education (IDOR), Rio de Janeiro, Rio de Janeiro, Brazil